CLINICAL TRIAL: NCT05242055
Title: A Prospective, Cohort, and Observational Study of the Effect of Integrated Diagnosis and Treatment of Chronic Kidney Disease (CKD) on Clinical Outcomes in Real World Clinical Practice
Brief Title: Integrated Diagnosis and Treatment of CKD on Outcomes
Status: Recruiting | Type: Observational
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Dongliang Zhang, MD, Director of Nephrology Department of Beijing Jishuitan Hospital, Peking University
Other Study IDs: 202112-11
Record Dates: First submitted 2022-01-29; First posted 2022-02-16 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Chronic Kidney Diseases; Hypertension; Hyperglycemia; Hyperlipidemias; Anemia; Chronic Kidney Disease-Mineral and Bone Disorder; Malnutrition
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension; Hyperglycemia; Hyperlipidemias; Anemia; Chronic Kidney Disease-Mineral and Bone Disorder; Malnutrition | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Integrated group: Patients in the integrated group should be the patients getting integrated diagnosis and treatment during following up period. Integrated diagnosis and treatment includes control of hypertension, hyperglycemia, hyperlipidemia, anemia, CKD-MBD, and malnutrition by regular follow-up according to the guidelines of Kidney Disease- Improving Global Outcomes and of Chinese Medical Association in 2021.
  Interventions: Other: Integrated diagnosis and treatment for CKD
- Unintegrated group: Patients in the unintegrated group are those who do not follow the contents of guidelines in some items of the integrated diagnosis and treatment during follow-up.
  Interventions: Other: Integrated diagnosis and treatment for CKD

INTERVENTIONS:
Other: Integrated diagnosis and treatment for CKD — This is an observational study. Investor will not intervene the clinical practice of doctors. In the real world, there would be many factors affect the proceeding of the guidelines contents. There will be integrated diagnosis and treatment during follow-up.

SUMMARY:
Objective: To establish a study cohort and follow up of patients with CKD in our hospital, and evaluate the status of integrated CKD diagnosis and treatment according to guidelines in the real world, as well as the clinical prognosis of patients with different stratification.

Methods: By establishing a cohort of 1000 patients with CKD and conducting long-term follow-up, integrated diagnosis and treatment for CKD was performed, namely: Regular monitoring, control of blood pressure, blood glucose, blood lipid, correction of anemia, minerals - bone metabolic abnormalities, malnutrition, acid and alkali, and electrolyte disorder, diet and exercise, such as the guidance of integrated management, non intrusive, observational studies, prospective cohort were analyzed retrospectively, describe the implementation of the integration of diagnosis and treatment, chronic kidney disease (CKD) Stratified analysis and risk factor analysis were performed for cardiovascular disease and other main endpoint events, so as to objectively reflect the status of integrated treatment of CKD and provide data support for continuous quality improvement of CKD diagnosis and treatment and improvement of clinical prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old;
* Voluntarily signed informed consent;
* Patients who are estimated to develop CKD.

Exclusion Criteria:

* Age < 18 or ≥100 years;
* Unable to comply with the procedures stipulated in this study;
* Estimated follow-up time ≤6 months.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CKD following up more than 6 months in Beijing Jishuitan Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of cardiovascular cerebrovascular adverse events | Six months or more
  Acute myocardial infarction, heart failure, shock, cardiac arrest, stroke, and lower limb arterial occlusion occurred during follow-up

SECONDARY OUTCOMES:
Rate of all-cause mortality | Six months or more
  Deaths from all causes during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Nephrology Department of Beijing Jishuitan Hospital, Beijing, Beijing Municipality, China